CLINICAL TRIAL: NCT04039529
Title: Novel Guidance Device for Image Fusion and Needle Guidance in Lung, Liver or Kidney Biopsy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: covid pandemic
Sponsor: Clear Guide Medical (Industry)
Collaborators: Temple University (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TUH SCENERGY
Record Dates: First submitted 2019-07-29; First posted 2019-07-31 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Liver Biopsy; Lung Biopsy; Kidney Biopsy
Keywords: lung biopsy; kidney biopsy; liver biopsy; image fusion

STUDY DESIGN:
Intervention Model Description: testing whether biopsies and ablations performed with the SCENERGY result in less patient radiation dose or reduced procedure time compared to biopsies performed under CT-guidance only.
Masking Description: Masking is impossible due to the hardware that is present when using the SCENERGY
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- CT-only guided biopsy (No Intervention): The current standard of care for biopsy at Temple University Hospital.
- SCENERGY-guided Biopsy (Experimental): The use of the SCENERGY to fuse CT and Ultrasound for biopsy
  Interventions: Device: SCENERGY-guided Biopsy

INTERVENTIONS:
Device: SCENERGY-guided Biopsy — Use of SCENERGY during a lung, liver or kidney biopsy
  Arms: SCENERGY-guided Biopsy

SUMMARY:
This study investigates whether a new image fusion technology can reduce patient radiation dose from CTs and/or procedure time during biopsies of lung, liver or kidney.

DETAILED DESCRIPTION:
This study proposes the use of a new fusion technology, Scenergy (Clear Guide Medical; FDA 510(k) K171677), which fuses CT images to real-time US images to minimize the drawbacks of each modality while enhancing their benefits. Such benefits include, the reduction of radiation dose to the patient with the fusion of initial CT imaging overlaying the live US images. The fused imaging software allows the operator to watch the needle tip advance towards the lesion on both live US and overlaid CT imaging. In such a setting, the operator would only need to perform an initial CT scan, advance the needle into position using fused US/CT images, and a final CT scan to ensure needle tip location. This eliminates interval CT scans that are usually required after each incremental needle position adjustment, and thus, reduces radiation dose to the patient and wasted procedural time during the incremental CT scans.

ELIGIBILITY:
Inclusion Criteria:

* all patients between the ages of 18 and 80 years old at time of procedure who are pre-scheduled for a lung, kidney, or liver biopsy.

Exclusion Criteria:

* any patient who was under the age of 18 or over the age of 80 at time of the procedure or who does not wish to volunteer for the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12-31 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Radiation Dose during Procedure | 1 hour
  The number of CTs or Fluoroscopy shots during the biopsy

SECONDARY OUTCOMES:
Time to Reach Target of Biopsy | 1 hour
  The amount of time in seconds that the physician takes to reach the target of biopsy
Experience Level | 1 hour
  Number of years physician has practiced in Interventional Radiology

CONTACTS AND LOCATIONS:
Locations (1):
- Temple University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No